CLINICAL TRIAL: NCT02301091
Title: Combine Transcatheter Arterial Embolization and Radiofrequency Ablation Versus Transcatheter Arterial Embolization Alone for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: Combine TACE and RFA Versus TACE Alone for HCC With PVTT
Acronym: CORTT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ming Zhao (Other)
Responsible Party: Sponsor-Investigator, Ming Zhao, Chief physician in Minimally Invasive Interventional Division,Medical Imaging Center,Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-FXY-036
Record Dates: First submitted 2014-11-13; First posted 2014-11-25 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC PVTT TACE RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic; pirarubicin; Mitomycin; lobaplatin; Cytotoxins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE-RFA (Experimental): 2 times TACE first, RFA for residual viable tumors and PVTT within 1 month.
  Interventions: Procedure: TACE; Procedure: RFA; Drug: pirarubicin,mitomycin and lobaplatin
- TACE alone (Active Comparator): repeated TACE and 1 to 2 months interval between two sessions of TACE.
  Interventions: Procedure: TACE; Drug: pirarubicin,mitomycin and lobaplatin

INTERVENTIONS:
Procedure: TACE — TACE will be done according to the current method in our center. We use intra-injection of lipiodol mixed with pirarubicin,mitomycin and lobaplatin when the catheter was placed in the superselective location very close to the tumor. Gelfoam sponge was then injected to temporarily occlude the arterial blood flow.
  Other Names: Transcatheter Arterial Chemoembolization; Chemoembolization
Procedure: RFA — For RFA, we used two commercially available system (Cool-Tip, Valleylab，USA) and (Octopus RF Systema，Starmed,Korea）with needle electrode with a 17-gauge internally cooled electrode.
  Other Names: Radiofrenquency ablation; RF ablation
  Arms: TACE-RFA
Drug: pirarubicin,mitomycin and lobaplatin — They were cytotoxic drugs used in the TACE procedure.
  Other Names: cytotoxic drugs

SUMMARY:
The purpose of this study is to determine whether combined radiofrequency ablation and transcatheter chemoembolization (TACE) result in better survival outcomes than TACE alone in patients with HCC and portal vein tumor thrombus.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the second most common cause of death from cancer globally. Although the development of imaging techniques has improved early HCC diagnosis, portal vein tumor thrombus (PVTT) is still identified in 12.5-39.7% of HCC patients at their initial visits. Patients suffering from extremely aggressive HCC with PVTT have a median survival time of only 2.7-4.0 months if left untreated. The current standard of practice recommends sorafenib, which has been shown to prolong overall survival (OS) by nearly 3 months in advanced HCC patients and by 1.5-3.2 months in those with PVTT.

Transarterial chemoembolization (TACE) is the main treatment modality for unresectable HCC patients. Some recent prospective studies have demonstrated that TACE can serve as a safe and effective procedure in selected HCC patients with PVTT. TACE is recommend for a part of patients with HCC and PVTT by the treatment guidelines in China and Japan. However,due to the poor blood supplement of PVTT,the local control rate of PVTT after TACE treatment is low. Besides,as to some hypovascular intrahepatic tumors, TACE also could not controlled effectively. As regard to the high local control rate of radiofrequency ablation (RFA) for intrahepatic lesions and PVTT reported in some studies, we thus suggested that the combination of TACE and RFA might have higher tumor control rate and survival benefit than TACE alone.

We design this study to compare survival outcomes of TACE plus RFA and TACE alone in patients with HCC and PVTT.A total of 240 patients are needed according to statistician's calculation.They will be divided into two groups randomly by computer after sign the informed consent form.One group of patients received TACE plus RFA and the other group of patients received TACE alone.After treatment,patients will be followed-up on their survival, tumor response and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* HCC with portal vein tumor thrombus in the first or second branch
* Refused sorafenib or could not tolerate the adverse effect of sorafenib
* A solitary HCC ≤ 5.0 cm in diameter, or multiple HCC ≤ 3 lesions, each ≤ 5.0 cm in diameter
* Eastern Cooperative Oncology Group Performance Status 0-1
* Child-Pugh Score ≤ 8
* A platelet counts of > 60,000/mm3, hemoglobin>8.5 g/dL, prothrombin time prolong <6s
* Albumin >2.8 g/dL, total bilirubin <51.3 umol/L; alanine aminotransferase (ALT) and aspartate transaminase（AST）<5 times of upper limit
* Sign the informed consent.

Exclusion Criteria:

* Presence of extrahepatic metastasis except lymph node metastasis
* The blood supply of tumor lesions is absolutely poor or arterial-venous shunt that TACE can not be performed
* Uncontrolled or refractory ascites, ongoing variceal bleeding or encephalopathy;
* Severe heart, brain or kidney diseases
* Previous or concurrent cancer that is distinct in primary site or histology from HCC
* Pregnant women or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival rates | 1 year

SECONDARY OUTCOMES:
Progression-free survival rates | 6 months
Response rate of PVTT | 6 months
Number of participants with adverse events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Minimally Invasive Interventional Division, Medical Imaging Center, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China